CLINICAL TRIAL: NCT01031927
Title: Sarcosine as Primary or Adjunctive Therapy in Obsessive Compulsive Disorder: A Prospective, Open-label Study
Brief Title: N-methyl Glycine (Sarcosine) for the Treatment of Obsessive Compulsive Disorder (OCD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Taipei City Hospital (Other Government)
Responsible Party: Po-Lun Wu, China Medical University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMR96-IRB-75
Record Dates: First submitted 2009-12-13; First posted 2009-12-15 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-12

CONDITIONS: Obsessive Compulsive Disorder
Keywords: obsessive compulsive disorder; sarcosine; glycine transporter I; NMDA receptor
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Sarcosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: N-methyl glycine — staring from 500mg/day, increased by 500mg biweekly, up to maximin of 2000mg/day
  Other Names: sarcosine

SUMMARY:
Several lines of evidence implicate glutamatergic dysfunction in the pathophysiology of obsessive compulsive disorder (OCD). Sarcosine, also known as N-methylglycine, is an endogenous antagonist of glycine transporter-I (GlyT-I), which potentiates glycine's action at the glycine site of N-methyl-D-aspartate (NMDA) receptors. In this 10-week open-label trial, we examined the efficacy and safety of sarcosine treatment in OCD patients.

ELIGIBILITY:
Inclusion Criteria:

* a primary OCD according to DSM-IV
* at least 1 year's duration of OC symptoms and a minimum severity score of ≥16 on Yale-Brown Obsessive Compulsive Scale
* drug naïve at study entry or
* being free from psychotropic medication for at least 8 weeks at study entry,or
* inadequately responded to ongoing psychotropic medications at study entry (defined by a Y-BOCS score of ≧16 despite treatment with maximum tolerated dose of a SRI medication for at least 8 weeks)

Exclusion Criteria:

* patients with moderate to severe depression defined by a 21-item Hamilton Depression Rating Scale score of >17,
* a history of bipolar disorder, schizophrenia, schizoaffective disorder, or other psychosis as defined by DSM-IV, or if they were at significant risk of suicide, and
* with clinically significant organic disease including cardiovascular, hepatic, pulmonary, neurologic, metabolic, or renal disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale | week0, 2, 4, 6, 8, and 10

SECONDARY OUTCOMES:
Hamilton Anxiety Rating scale | week0, 2, 4, 6, 8, and 10

CONTACTS AND LOCATIONS:
Overall Officials: Guochuan E Tsai, MD, PhD, Study Chair — Department of Psychiatry, Harbor-UCLA Medical Center, California, U.S.A
Locations (1):
- China Medical University Hospital, Taichung, Taiwan